CLINICAL TRIAL: NCT03259360
Title: A Facebook Intervention for Young Sexual and Gender Minority Smokers
Acronym: POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-15-263; R21MD011765 (NIH); K23DA032578 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use; Smoking; Tobacco Dependence; Tobacco Use Disorder; Tobacco Use Cessation; Tobacco Smoking; Smoking Cessation; Smoking, Cigarette; Smoking, Tobacco
Keywords: Tobacco; Gender Identity Minority; Sexual Identity Minority; Cessation; Intervention; Young Adults; Social Media; Internet; Cigarette
MeSH Terms: conditions — Tobacco Use; Smoking; Tobacco Use Disorder; Tobacco Use Cessation; Tobacco Smoking; Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Put It Out Project (POP): (Experimental): a culturally tailored intervention developed for SGM young adults on Facebook
  Interventions: Behavioral: POP:
- Tobacco Status Project (TSP): (Experimental): the original TSP intervention (non-tailored) delivered to groups of only SGM participants on Facebook
  Interventions: Behavioral: TSP:

INTERVENTIONS:
Behavioral: POP: — 90 days of Facebook messaging, weekly live sessions targeting tobacco use and tailored to sexual and gender minority young adults
  Arms: The Put It Out Project (POP):
Behavioral: TSP: — 90 days of Facebook messaging, weekly live sessions targeting tobacco use
  Arms: Tobacco Status Project (TSP):

SUMMARY:
The 2-year research plan will test the Put It Out Project (POP) in a pilot randomized trial (N=120) compared to TSP and two historical control conditions. Participants will be young adults who smoke, identify as sexual or gender minorities, and use Facebook. The primary outcome will be biochemically verified 7-day abstinence from smoking at 3 and 6 months. Secondary outcomes will be a quit attempt (y/n), stage of change, and thoughts about tobacco abstinence at 3 and 6 mos.

DETAILED DESCRIPTION:
Participants will be randomized to one of two conditions: (1) a Facebook-delivered intervention addressing tobacco use, tailored to SGM young adults; or (2) a 3-month Facebook intervention targeting tobacco use. Both interventions will include 90 days of Facebook-based messages and activities tailored to participants' readiness to quit smoking.

Assessments will occur at baseline, 3, and 6 months follow-up. Assessments will include measures on smoking, thoughts about abstinence, and SGM identity experiences. All participants who report no past 7-day smoking will be asked to give biochemical verification of smoking status with saliva cotinine test kits that will be mailed to participants.

ELIGIBILITY:
Inclusion Criteria:

* read English
* between 18 and 25 years of age
* indicate they use Facebook "most" (≥ 4) days per week
* have smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* identifies as SGM

Exclusion Criteria:

* do not read English
* are not between 18 and 25 years of age
* indicate they do not use Facebook "most" (≥ 4) days per week
* have not smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* does not identify as SGM

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence at 3 months | 3 months post baseline
  Reports of no smoking in the 7 days prior to the 3 month assessment. Biochemical verification of abstinence will also be recorded.
7-day point prevalence abstinence at 6 months | 6 months post baseline
  Reports of no smoking in the 7 days prior to the 6 month assessment. Biochemical verification of abstinence will also be recorded.

SECONDARY OUTCOMES:
Reduction in cigarettes smoked by at least 50% | 3 and 6 months post baseline
  Reduction will be assessed at 3 and 6 month follow-ups.
Tobacco use quit attempts | 3 and 6 months post baseline
  Whether a quit attempt was made during the follow-up period at 3 and 6 months post-baseline.
Readiness to quit tobacco | 3 and 6 months post baseline
  Proportion of participants ready to quit smoking in the next month assessed at 3 and 6 months
Thoughts About Tobacco Abstinence | 3 and 6 months post baseline
  Desire to quit, abstinence self-efficacy, perceived difficulty of quitting and abstinence goal

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Humfleet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Department of Psychiatry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramo DE, Thrul J, Chavez K, Delucchi KL, Prochaska JJ. Feasibility and Quit Rates of the Tobacco Status Project: A Facebook Smoking Cessation Intervention for Young Adults. J Med Internet Res. 2015 Dec 31;17(12):e291. doi: 10.2196/jmir.5209. PMID 26721211
- [Background] Thrul J, Klein AB, Ramo DE. Smoking Cessation Intervention on Facebook: Which Content Generates the Best Engagement? J Med Internet Res. 2015 Nov 11;17(11):e244. doi: 10.2196/jmir.4575. PMID 26561529
- [Background] Ramo DE, Thrul J, Delucchi KL, Ling PM, Hall SM, Prochaska JJ. The Tobacco Status Project (TSP): Study protocol for a randomized controlled trial of a Facebook smoking cessation intervention for young adults. BMC Public Health. 2015 Sep 15;15:897. doi: 10.1186/s12889-015-2217-0. PMID 26374203
- [Background] Ramo DE, Rodriguez TM, Chavez K, Sommer MJ, Prochaska JJ. Facebook Recruitment of Young Adult Smokers for a Cessation Trial: Methods, Metrics, and Lessons Learned. Internet Interv. 2014 Apr;1(2):58-64. doi: 10.1016/j.invent.2014.05.001. PMID 25045624
- [Background] Ramo DE, Liu H, Prochaska JJ. A mixed-methods study of young adults' receptivity to using Facebook for smoking cessation: if you build it, will they come? Am J Health Promot. 2015 Mar-Apr;29(4):e126-35. doi: 10.4278/ajhp.130326-QUAL-128. Epub 2014 Feb 27. PMID 24575728
- [Background] Vogel EA, Ramo DE, Meacham MC, Prochaska JJ, Delucchi KL, Humfleet GL. The Put It Out Project (POP) Facebook Intervention for Young Sexual and Gender Minority Smokers: Outcomes of a Pilot, Randomized, Controlled Trial. Nicotine Tob Res. 2020 Aug 24;22(9):1614-1621. doi: 10.1093/ntr/ntz184. PMID 31562765

DOCUMENTS (1):
  • Informed Consent Form (2017-11-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03259360/ICF_000.pdf